CLINICAL TRIAL: NCT04030234
Title: Effects of Intensive Systolic Blood Pressure Lowering Treatment in Reducing RIsk of Vascular evenTs (ESPRIT) Study
Acronym: ESPRIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018YFC1312400
Record Dates: First submitted 2019-07-17; First posted 2019-07-23 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-01

CONDITIONS: Hypertension
Keywords: Hypertension; Blood pressure target
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive treatment group (Experimental): Participants randomized into the Intensive treatment group will have a goal of SBP <120 mmHg. A two- or three-drug regimen should be initiated at randomization for most participants. Drug doses should be increased and/or additional antihypertensive medications should be added at each visit in the intensive treatment group, usually at monthly intervals, until the participant's goal of <120 mmHg has been reached or the local investigator decides no further antihypertensive medications may be added.
  Interventions: Drug: Intensive BP treatment group
- Standard treatment group (Active Comparator): Participants randomized into the Standard treatment group will have a goal of SBP <140 mmHg. It is expected to achieve a SBP of 135-139 mmHg in as many participants as possible. Medication dose titration or addition of another drug is indicated if SBP is ≥160 mmHg at a single visit or is ≥140 mmHg at two consecutive visits. Down titration should be carried out if the SBP is <130 mmHg at a single visit or <135 mmHg at two consecutive visits.
  Interventions: Drug: Standard BP treatment group

INTERVENTIONS:
Drug: Intensive BP treatment group — Participants in the Intensive BP treatment group have a goal of SBP <120 mmHg. It is recommended to provide long-acting antihypertensive medications, that is once daily, unless other medication delivery frequency is needed. The local investigator may select among the available study antihypertensive medications. Other drugs not supplied by the trial may also be used as the investigator determines appropriate.
  One or more medications from the following classes of agents will be provided by the study for use in managing participants in both randomization groups to achieve study goals:
  Angiotension converting enzyme (ACE)-inhibitors; Angiotension receptor blockers (ARBs); Thiazide-type diuretics; Loop diuretics; Potassium-sparing diuretics; Beta-blockers; Calcium channel blockers (CCBs); Direct vasodilators; Alpha1-receptor blockers; Sympatholytics
  Other Names: Control of SBP to <120 mmHg
  Arms: Intensive treatment group
Drug: Standard BP treatment group — Participants in the Standard BP treatment group have a goal of SBP <140 mmHg. The same medications used in the Intensive BP treatment group will be used for the Standard BP treatment group.
  Other Names: Control of SBP to <140 mmHg
  Arms: Standard treatment group

SUMMARY:
This trial aims to assess, in patients aged ≥50 years with an average baseline SBP ≥130 mmHg and a previous history of cardiovascular diseases or at high vascular risk, the effects on the incidence of major cardiovascular events during the scheduled treatment period of greater reduction in blood pressure with a SBP target <120 mmHg versus <140 mmHg.

DETAILED DESCRIPTION:
This study is a multicenter, open-label, randomized controlled trial, which will randomize participants aged ≥50 years with an average baseline SBP ≥130 mmHg and a previous history of cardiovascular diseases or at high vascular risk. The study will compare the effects on the incidence of major cardiovascular events of allocation to achieve an intensive SBP goal (SBP <120 mmHg) with a standard SBP goal (SBP <140 mmHg) in four years of follow up.

ELIGIBILITY:
Inclusion Criteria:

1. At least ≥50 years old, and
2. Systolic blood pressure (SBP): (having documentation of SBP to meet the criteria below on 2 consecutive visits)

   * SBP: 130-180 mmHg on 0 or 1 medication
   * SBP: 130-170 mmHg on up to 2 medications
   * SBP: 130-160 mmHg on up to 3 medications
   * SBP: 130-150 mmHg on up to 4 medications, and
3. Prior vascular disease or at high vascular risk

   1. Previous myocardial infarction (MI), percutaneous coronary intervention (PCI), coronary artery bypass grafting (CABG), at least a 50% diameter stenosis of a coronary, chest pain with objective evidence of myocardial ischemia (load electrocardiogram or load image examination indicated myocardial ischemia)
   2. Previous stroke
   3. Carotid endarterectomy (CE), or carotid stenting
   4. Peripheral artery disease (PAD) with revascularization
   5. Abdominal aortic aneurysm (AAA) ≥5 cm with repair
   6. Combine with no less than two risk factors below

      * ≥60 years old male or ≥65 years old female
      * Diabetes
      * Dyslipidemia (total cholesterol >200 mg/dL [5.2 mmol/L] or LDL-C >130 mg/dL [3.4 mmol/L] or HDL-C < 40 mg/dL [1.0 mmol/L])
      * Current smoking (smoke more than a cigarette every day in the past 12 months)

Exclusion Criteria:

1. Known secondary cause of hypertension
2. An indication for a specific BP lowering medication that the participant is not taking and the participant has not been documented to be intolerant of the medication class
3. One minute standing SBP <110 mmHg (not applicable if unable to stand)
4. Arm circumference too large or small to allow accurate blood pressure measurement with available devices
5. Proteinuria defined as urine dipstick ≥2+ protein at screening
6. Glomerulonephritis treated with or likely to be treated with immunosuppressive therapy
7. eGFR <45 ml/min /1.73m2 or end-stage renal disease (ESRD)
8. Previous MI, stroke, or hospitalization for angina, PCI, CABG, CE or carotid stenting, PAD with revascularization, AAA≥5 cm with repair within last 3 months
9. Symptomatic heart failure within the past 6 months or documented left ventricular ejection fraction (by any method) <35%
10. PCI or CABG planned for the next 6 months
11. A medical condition likely to limit survival to less than 3 years, or a cancer (other than non-melanoma skin cancer) diagnosed and treated within the past two years that, in the judgment of local clinical investigators, would compromise a participant's ability to comply with the protocol and complete the trial
12. Any organ transplant
13. Pregnancy, breast-feeding, or of child-bearing potential and not using adequate contraception
14. Any factors judged by local clinic investigators to be likely to limit adherence to interventions. For example,

    1. Active alcohol or substance abuse within the last 12 months
    2. Plans to move to another place to live for a long time
    3. Clinical diagnosis of dementia or mild cognitive impairment (MCI)
15. Currently participation in a clinical trial with an unlicensed drug or device
16. Living in the same household as an already randomized participant

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11255 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
Number of participants with composite of major CVD events | 4 years
  Composite outcome of myocardial infarction, coronary or non-coronary revascularization, chronic or acute decompensated heart failure hospitalization or emergency department visit, stroke, or death from cardiovascular disease

SECONDARY OUTCOMES:
Number of participants with myocardial infarction | 4 years
Number of participants with coronary revascularization | 4 years
Number of participants with non-coronary revascularization | 4 years
Number of participants with chronic or acute decompensated heart failure hospitalization or emergency department visit | 4 years
Number of participants with stroke | 4 years
Number of participants with cardiovascular death | 4 years
Number of participants with all-cause death | 4 years
Number of participants with composite outcome of the primary composite with all-cause death | 4 years
Number of participants with end-stage kidney disease (ESKD), a sustained decline in eGFR to <10 mL/min/1.73m2, renal death, or a sustained decline of ≥40% in eGFR from randomization | 4 years
Number of participants with all-cause dementia or mild cognitive impairment | 4 years
Difference of arteriole-to-venule ratio measured by fundus photography between intensive treatment group and standard treatment group | at 4-year final follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Jing Li, MD, PhD, Principal Investigator — National Center for Cardiovascular Diseases; Jiamin Liu, MD, Principal Investigator — National Center for Cardiovascular Diseases
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Huang X, Zhang H, Li Y, Ge J, Sun Y, Zhang L, Zhao L, Liu J, Zhang C, Du J, Li Y, Zhang H, Hao F, Wang Q, Xu W, Liu J, Li J. Modest Effects of Intensive Blood Pressure-Lowering on Quality of Life in Patients at High Cardiovascular Risk: The ESPRIT Trial. J Am Coll Cardiol. 2025 Oct 28;86(17):1392-1401. doi: 10.1016/j.jacc.2025.06.010. Epub 2025 Oct 17. PMID 41105075
- [Derived] Wang B, Shi D, Zhang Z, Zhang L, Sun Y, Liu J, Yan X, Jing J, Li J, Song J, Li Y, Li G, Zhang L, Wang Z, Chen J, Zhang W, Cai S, Han S, Luan T, Yi S, Su S, Du J, Kou X, Liu J, Dai X, Li N, Zhu J, Tang C, Liu S, Su H, Liu Y, Mao Y, Yang X, He M, Zhang Q, Li J. Effect of Intensive Blood Pressure Lowering Treatment on Retinal Microvasculature: Secondary Analysis From ESPRIT. J Am Coll Cardiol. 2025 Oct 28;86(17):1377-1388. doi: 10.1016/j.jacc.2025.05.020. Epub 2025 Oct 17. PMID 41105073
- [Derived] Li S, Peng Y, Li Y, Sun Y, Yan X, Zhang L, Liu J, Zhao L, Liu J, Qian J, Zhai N, Dong L, Ruan J, Zhang P, Wei X, Liu Y, Ma Q, Huang W, Zhang Q, An C, Liu J, Sheng L, Zhang H, Li J; ESPRIT Investigators. Effects of Intensive Blood Pressure Control in Patients With Frailty: A Post Hoc Analysis From ESPRIT. J Am Coll Cardiol. 2026 Jan 6;87(1):4-16. doi: 10.1016/j.jacc.2025.08.092. Epub 2025 Oct 15. PMID 41091084
- [Derived] Liu J, Li Y, Ge J, Yan X, Zhang H, Zheng X, Lu J, Li X, Gao Y, Lei L, Liu J, Li J; ESPRIT Collaborative Group. Lowering systolic blood pressure to less than 120 mm Hg versus less than 140 mm Hg in patients with high cardiovascular risk with and without diabetes or previous stroke: an open-label, blinded-outcome, randomised trial. Lancet. 2024 Jul 20;404(10449):245-255. doi: 10.1016/S0140-6736(24)01028-6. Epub 2024 Jun 27. PMID 38945140
- [Derived] Saiz LC, Gorricho J, Garjon J, Celaya MC, Erviti J, Leache L. Blood pressure targets for the treatment of people with hypertension and cardiovascular disease. Cochrane Database Syst Rev. 2022 Nov 18;11(11):CD010315. doi: 10.1002/14651858.CD010315.pub5. PMID 36398903
- [Derived] Saiz LC, Gorricho J, Garjon J, Celaya MC, Erviti J, Leache L. Blood pressure targets for the treatment of people with hypertension and cardiovascular disease. Cochrane Database Syst Rev. 2020 Sep 9;9(9):CD010315. doi: 10.1002/14651858.CD010315.pub4. PMID 32905623